CLINICAL TRIAL: NCT01393535
Title: Study of the Relationship Between Serum Adiponectin and Clinical Prognosis in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Chunhu Gu, Xijing Hospital
Other Study IDs: Guch-013
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Cardiac Surgery
Keywords: Adiponectin; Prognosis; Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the relationship between serum adiponectin and clinical prognosis in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Adiponectin, an adipose tissue derived protein, is an abundant protein hormone regulatory of numerous metabolic processes. Since its discovery, adiponectin has garnered considerable attention for its role in cardiovascular pathology. It has been shown to be a predictor of cardiovascular events in both the general population and patients undergoing cardiac surgery. In this study,we are planning to investigate the relationship between serum adiponectin and clinical prognosis in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had underwent cardiac surgery from July 2011 to August 2012 in xijing hospital.

Exclusion Criteria:

* Nothing particular.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent cardiac surgery in cardiovascular surgery department of xijing hospital.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dinghua Yi, MD, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China